CLINICAL TRIAL: NCT04400695
Title: Randomized, Controlled, Multicenter Phase III Clinical Study Evaluating the Efficacy and Safety of RC48-ADC for the Treatment of Locally Advanced or Metastatic Breast Cancer With Low Expression of HER2
Brief Title: A Study of RC48-ADC for the Treatment of Locally Advanced or Metastatic Breast Cancer With Low Expression of HER2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C012
Record Dates: First submitted 2020-04-30; First posted 2020-05-22 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Docetaxel; Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC48-ADC (Experimental): RC48-ADC common name：Recombinant Humanized anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection Dosage form：Lyophilized powder injection specification：60 mg / piece Medication plan：Every 2 weeks Expiration date：18 months HER2-low, unresectable, locally advanced or metastatic breast cancer participants previously treated with anthracycline and received 1 or 2 systemic chemotherapy after relapse / metastasis.
  Interventions: Drug: RC48-ADC
- Physician's Choice (Active Comparator): Physician's Choice:
  HER2-low, unresectable, locally advanced or metastatic breast cancer participants previously treated with anthracycline and received 1 or 2 systemic chemotherapy after relapse / metastasis.
  Physician's choice from the following options:
  Paclitaxel Injection Docetaxel Injection Vinorelbine Tartrate Injection Capecitabine Tablets
  Interventions: Drug: Paclitaxel Injection; Drug: Docetaxel Injection; Drug: Vinorelbine Tartrate Injection; Drug: Capecitabine Tablets

INTERVENTIONS:
Drug: RC48-ADC — RC48-ADC 2.0mg / kg, intravenous drip, once every 2 weeks
  Other Names: RC48
  Arms: RC48-ADC
Drug: Paclitaxel Injection — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Other Names: Taxol
  Arms: Physician's Choice
Drug: Docetaxel Injection — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Other Names: Taxotere
  Arms: Physician's Choice
Drug: Vinorelbine Tartrate Injection — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Other Names: Navelbine
  Arms: Physician's Choice
Drug: Capecitabine Tablets — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Other Names: Xeloda
  Arms: Physician's Choice

SUMMARY:
This study will compare RC48-ADC to physician choice standard treatment. Participants must have HER2-low breast cancer ，previous use of anthracyclines, and have been treated with one or two systemic chemotherapy regimens following recurrence/metastasis.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, open, parallel control to evaluate the effectiveness and safety of Phase III clinical trials of the efficacy and safety of recombinant humanized anti-HER2 monoclonal antibody-Monomethyl auristatin E (MMAE) conjugate for the treatment of locally advanced or metastatic breast cancer the study.The low expression of HER2 is defined as: the immunohistochemistry (IHC) confirmed by the central laboratory detects the expression of HER2 protein as IHC 2+ and the fluorescence in situ hybridization (FISH) detection has no amplification.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the study and sign the informed consent;
* Subjects aged 18-70 years (including 18 years and 70 years) and not reaching the 71st birthday were all considered to be ≤70 years old;
* Expected survival ≥12 weeks;
* Eastern Cooperative Oncology Group(ECOG) physical condition 0 or 1;
* For female subjects of child-bearing age women agreed to study during treatment and experimental subjects within 6 months after the end of the treatment period using an approved by the medical contraception (e.g. intrauterine device, the pill or condoms), before the study drug delivery within 7 days of pregnancy blood test must be negative (sterilization surgery or age 60 or more subjects can choose no pregnancy blood test), and must be an lactation. For male subjects: should be sterilized surgically, or agree to use a medically approved contraceptive method during the study period and for 6 months after the end of the treatment period. Control subjects after the end of the treatment period according to the choice of control drugs to determine the length of contraception.
* Able to understand the study requirements and be willing and able to follow the study and follow-up procedures.
* Bone marrow function:

hemoglobin ≥9g/dL; absolute neutrophil count ≥1.5×109/L; white blood cell count ≥3.0×109/L platelet ≥100 ×109/L;

* Liver function (according to the normal value of the clinical trial center) :

serum total bilirubin ≤1.5 times the upper limit of normal value (ULN); alanine aminotransferase (ALT), aspartate aminotransferase(AST) and Alkaline phosphatase（ALP） were ≤2.5 × ULN in the absence of liver metastasis, and ALT, AST and Alkaline phosphatase(ALP) were ≤5 × ULN in the presence of liver metastasis

* Renal function (according to the normal value of the clinical trial center) :

serum creatinine ≤1.5×ULN, or calculated by Cockcroft-Gault formula, the creatinine clearance rate (CrCl) ≥60 mL/min;

* Cardiac function:

American New York college of cardiology (NYHA) grade < 3; left ventricular ejection fraction ≥50%;

* Breast cancer subjects diagnosed by histology and / or cytology are currently at a locally advanced or metastatic stage and cannot be radically removed;
* The low expression of HER2 confirmed by the IHC and FISH results of the central laboratory (defined as: IHC 2+ and no amplification of FISH); the subject can provide a specimen of the primary or metastatic tumor site (paraffin wax) for HER2 detection Block, paraffin-embedded section or fresh tissue section can be used);
* Previous use of anthracycline drugs;
* Received 1 or 2 systemic chemotherapy treatments after relapse / metastasis. Subjects who relapsed during adjuvant chemotherapy or within 12 months after the end of adjuvant chemotherapy were considered to have failed first-line chemotherapy after relapse / metastasis.
* Hormone receptors are negative or positive. Hormone receptor-positive subjects need to progress after receiving endocrine therapy after relapse / metastasis or relapse after less than 2 years. Patients who are not suitable for endocrine therapy can be included in this study after undergoing chemotherapy treatment (first-line or second-line);
* The imaging evidence confirmed by the investigator that the tumor disease progressed during or after the most recent treatment is required;
* There has been no diagnosis of HER2 positive (HER2 IHC 3+ or FISH amplification)
* Have not used drugs targeting HER2 (including antibodies, small molecule Tyrosine kinase inhibitor（TKIs） and antibody drug conjugates).
* According to the RECIST 1.1 standard, there is at least one measurable lesion.

Exclusion Criteria:

* Received chemotherapy within 4 weeks before the start of study administration (treatment with nitrosourea and mitomycin C within 6 weeks, oral fluorouracil within 2 weeks), radiotherapy (palliative for bone metastases Local radiotherapy is within 2 weeks before study administration), immunotherapy; received endocrine therapy for breast cancer within 2 weeks before study administration;
* The research drug was used within 4 weeks before the start of study administration;
* Have undergone major surgery within 4 weeks before the start of study administration;
* Have received a live vaccine within 4 weeks before the start of study administration or plan to receive any vaccine during the study period;
* Serious cardiovascular and cerebrovascular events occurred within 12 months, including but not limited to unstable angina, myocardial infarction, cerebral hemorrhage, and cerebral infarction (except for asymptomatic and untreated lacunar infarction)；
* Those who are suffering from heart disease are not suitable for enrollment, including but not limited to arrhythmia and heart failure requiring medical treatment or accompanied by symptoms;
* There are other lung diseases requiring treatment or serious, including but not limited to active pulmonary tuberculosis, interstitial lung disease, etc ;
* Suffering from active infection requiring systemic treatment;
* Have active autoimmune diseases (such as the use of corticosteroids or immunosuppressive drugs, etc.) that require systemic treatment within the past 2 years, allowing related alternative treatments (such as thyroxine, insulin, or the physiology of adrenal or pituitary insufficiency Corticosteroid replacement therapy);
* The toxicity of the previous anti-tumor therapy has not been restored to the 0 to 1 level defined by CTCAE version 5.0, of which the neurotoxicity has not been restored to 0; except for hair loss, pigmentation or other researches that do not increase the risk of medication Happening;
* Have a clear past or current history of neurological or mental disorders, including epilepsy or dementia;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subject or affect the completion of the clinical study；
* Positive HIV test results; patients with active hepatitis B or C (HBsAg positive and hepatitis B virus（HBV） DNA titers above the upper limit of normal; Hepatitis C Virus Antibody(HCVAb) positive hepatitis C virus （HCV） RNA titers above the upper limit of normal)；
* There is a third interstitial fluid that cannot be controlled by drainage or other methods (including a large amount of pleural effusion or ascites);
* Known hypersensitivity or delayed allergic reaction to certain components of RC48-ADC or similar drugs;
* Subjects who are not suitable for using any of the alternative control drugs;
* The presence of brain metastases and / or cancerous meningitis;
* Have other malignant tumors within 5 years before signing the informed consent form (except for non-melanoma skin cancer, cervical carcinoma in situ or other tumors that have been effectively treated, except malignant tumors that are considered cured);
* Subjects who are estimated to be inadequate for patients to participate in this clinical study or other factors that the investigator believes are inappropriate to participate in this study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS), evaluated by an independent efficacy evaluation committee | within approximately 3 years
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard.

SECONDARY OUTCOMES:
Progression-free survival (PFS), evaluated by the investigator | within approximately 3 years
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard.
Objective remission rate (ORR) | within approximately 3 years
  The objective response rate will be mainly analyzed by the independent efficacy evaluation committee according to the RECIST 1.1 standard tumor evaluation (the evaluation by the investigator will also be performed).
Duration of relief (DOR) | within approximately 3 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death
Disease control rate (DCR) | within approximately 3 years
  Disease control rate (DCR) is defined as cases where objective remission (assessed as complete remission or partial remission according to RECIST 1.1 standard) or stable disease during the study.
Tumor progression time (TTP) | within approximately 3 years
  Time to disease progression (TTP) refers to the time from the random date to the first disease progression (calculated by the event that occurred first). Disease progression will be evaluated by the investigator according to the RECIST 1.1 standard (investigator and Independent Review Committee(IRC) evaluation).
Overall survival (OS) | within approximately 3 years
  Overall survival (OS) refers to the time from the date of randomization to the date of death of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Oncology Hospital, Chinese Academy of Medical Sciences; Tao Sun, Principal Investigator — Liaoning Cancer Hospital & Institute; Wei Li, Principal Investigator — Jilin University First Hospital; Yuee Teng, Principal Investigator — First Affiliated Hospital of China Medical University; Shu Wang, Principal Investigator — Peking University People's Hospital; Xiaojia Wang, Principal Investigator — Zhejiang Cancer Hospital; Min Yan, Principal Investigator — Henan Cancer Hospital; Jifeng Feng, Principal Investigator — Jiangsu Cancer Institute & Hospital; Ying Cheng, Principal Investigator — Jilin Provincial Tumor Hospital; Ying Wang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Ying Wang, Principal Investigator — Sun Yat-sen University Cancer Prevention and Control Center; Ning Liao, Principal Investigator — Guangdong Provincial People's Hospital; Haibo Wang, Principal Investigator — Qingdao University Hospital; Quchang Ouyang, Principal Investigator — Hunan Cancer Hospital; Yueyin Pan, Principal Investigator — Anhui Provincial Hospital; Yingying Du, Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Changlu Hu, Principal Investigator — Anhui Provincial Cancer Hospital; Zhongsheng Tong, Principal Investigator — Tianjin Cancer Hospital; Jin Yang, Principal Investigator — The First Affiliated Hospital of Xi'an Jiaotong University School of Medicine; Lihua Song, Principal Investigator — Shandong Cancer Hospital and Institute; Xiuwen Wang, Principal Investigator — Qilu Hospital of Shandong University; Yu Jiang, Principal Investigator — West China Hospital; Yunjiang Liu, Principal Investigator — Hebei Medical University Fourth Hospital; Jing Cheng, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Huihua Xiong, Principal Investigator — Tongji Hospital; Xinhong Wu, Principal Investigator — Hubei Cancer Hospital; Peng Shen, Principal Investigator — Zhejiang University; Weimin Xie, Principal Investigator — Cancer Hospital Affiliated to Guangxi Medical University; Xin Zhou, Principal Investigator — Chongqing University Cancer Hospital; Li Ran, Principal Investigator — Cancer Hospital of Guizhou Province; Yu Wang, Principal Investigator — Shanxi Province Cancer Hospital; Jinnan Gao, Principal Investigator — Bethune Hospital of Shanxi Province; Jingfen Wang, Principal Investigator — Linyi Cancer Hospital; Liangming Zhang, Principal Investigator — Yantai Yuhuangding Hospital; Xianhe Xie, Principal Investigator — First Affiliated Hospital of Fujian Medical University; Ru Zeng, Principal Investigator — The First Affiliated Hospital of Xiamen University; Airong Wang, Principal Investigator — Weihai Municipal Hospital; Zhengqiu Zhu, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Sanyuan Sun, Principal Investigator — Xuzhou Central Hospital; Qingshan Li, Principal Investigator — Affiliated Hospital of Chengde Medical College; Aimin Zang, Principal Investigator — Affiliated Hospital of Hebei University; Liuzhong Yang, Principal Investigator — The First Affiliated Hospital of Xinxiang Medical College; Meili Sun, Principal Investigator — Jinan Central Hospital; Liang Li, Principal Investigator — Zibo Central Hospital; Guohua Yu, Principal Investigator — Weifang People's Hospital; Xujuan Wang, Principal Investigator — Neijiang Second People's Hospital
Locations (1):
- Oncology Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No